CLINICAL TRIAL: NCT00784173
Title: Middle and Inner Ear Malformation in Children With Velocardiofacial Syndrome
Status: Completed | Type: Observational
Sponsor: Pontificia Universidade Catolica de Sao Paulo (Other)
Responsible Party: Alfredo Tabith Junior, Pontificia Universidade Catolica de São Paulo
Other Study IDs: Unique protocol
Record Dates: First submitted 2008-10-31; First posted 2008-11-03 (Estimated); Last update posted 2008-11-03 (Estimated); Status verified 2008-10

CONDITIONS: Ear Malformations in the Velocardiofacial Syndrome
Keywords: Syndrome; Velocardiofacial; Middle ear; Inner ear; Malformation
MeSH Terms: conditions — Syndrome; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Middle and inner ear malformations on two boys with velocardiofacial syndrome are discussed.Special attention should be given to the presence of hearing loss due to middle and inner ear malformations, in addition to frequent conductive hearing loss regarding mastoid and middle ear inflammatory processes.

DETAILED DESCRIPTION:
Two boys with clinical signs of velocardiofacial syndrome, at ages of 4.7 and 6,7 years old are the subjects of this study.Audiological evaluation, including pure tone audiometry, tympanometry, acoustical reflex, and Computerized Tomography of temporal bones, and analyses of DNA sample with markers of 22q11 region were performed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with velocardiofacial syndrome

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children with velocardiofacial syndrome
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2007-01; Primary Completion 2007-03 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Tabith-Junior, MD, Principal Investigator — Pontificia Universidade Católica de São Paulo